CLINICAL TRIAL: NCT00328588
Title: LUCY: A Study for the Treatment of Non-Small Cell Lung Cancer (NSCLC) in Patients Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-006
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2008-01-02 (Estimated); Status verified 2007-12

CONDITIONS: Lung Cancer; Cancer of Lung; Cancer of the Lung; Non-Small Cell Lung Carcinoma; Carcinoma, Non-Small Cell Lung
Keywords: Treatment Efficacy; Treatment Effectiveness; Disease Management; Treatment; Safety
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — sepantronium

ARMS (1):
- 1 (Experimental): 7 days continuous infusion
  Interventions: Drug: YM155

INTERVENTIONS:
Drug: YM155 — IV

SUMMARY:
A study for the treatment of Non-Small Cell Lung Cancer (NSCLC) in patients previously treated with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer.
* Prior chemotherapy regimen(s) for lung cancer

Exclusion Criteria:

* History of other malignancy in the last 5 years
* Major surgery within the past 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Tumor response rate (CR+PR) | In first 6 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (6):
- Czechia (4):
  - Chomutov
  - Novi Jicin
  - Ostrava
  - Prague
- Großhansdorf, Germany
- Amsterdam, Netherlands